CLINICAL TRIAL: NCT05115656
Title: The Effectiveness and Underlying Mechanism of a Wellbeing Program for Traumatic Brain Injury - A Randomized Clinical Trial
Brief Title: Online Intervention for Traumatic Brain Injury Wellbeing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jean Lengenfelder, Assistant Director, Kessler Foundation
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R-1037-18; 90IFRE0016 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2021-10-20; First posted 2021-11-10 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury; Attention Impaired; Emotional Regulation
Keywords: Intervention; Psychological; Emotional; Well-being; Memory; Attention; Problem-Solving
MeSH Terms: conditions — Brain Injuries, Traumatic; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants (Moderate to Severe TBI patients) will be randomized into one of 2 online group interventions.
Who Masked: Participant, Investigator
Masking Description: Rigorous, Double-Masked/Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online group intervention 1 (Experimental): Participants in group 1 meet weekly online for a 2-hour group sessions for 10 weeks where the instructor will provide leadership in discussions, which will include practice of basic routines. Participants will also be asked to do 20-30 minutes of daily activities/exercises, where they will be asked to practice mental exercises.
  Interventions: Behavioral: Online group 1
- Online group intervention 2 (Active Comparator): Similar to group 1, participants will meet weekly online or in person for 2-hour group sessions for 10 weeks where the instructor will provide leadership in discussions, which will include practice of basic routines. Participants will also be asked to do 20-30 minutes of daily activities/exercises, where they will be asked to practice mental exercises.
  Interventions: Behavioral: Online group 2

INTERVENTIONS:
Behavioral: Online group 1 — The intervention is specifically tailored to meet particular cognitive standard and satisfy the needs of brain injury patients. For 2-3 hours weekly, participants will be immersed in mental exercises designed to help them overcome various challenges.
  Arms: Online group intervention 1
Behavioral: Online group 2 — The intervention is specifically tailored to meet particular cognitive standard and satisfy the needs of brain injury patients. For 2-3 hours weekly, participants will be immersed in mental exercises designed to help them overcome various challenges.
  Arms: Online group intervention 2

SUMMARY:
Traumatic brain injury (TBI) patients face notable impairments which lead to reduced performance and regulation of daily and overall functioning. There are a number of interventions made to combat these qualms; however, such interventions have historically been therapeutically demanding, which limits their practical benefit. An online therapeutic intervention can provide a cost-effective approach that can be particularly well-suited to the needs and limitations of TBI. It focuses both on developing awareness and attention, which are often impaired, and are critical to improving emotional and behavioral regulation and everyday function.

This project is aimed at assessing the effectiveness and underlying mechanism of modified mindfulness based stress reduction (MBSR) using a rigorous randomized controlled trial. Poised to provide a rigorous approach to efficacy development and analysis, Results of the study will provide valuable information that will ultimately support the refinement of an intervention that can have a real impact on patients' ability to resume a fully functional and satisfying life, and the design of an adequate therapeutic intervention for TBI patients.

DETAILED DESCRIPTION:
TBI patients suffer from a host of cognitive and behavioral deficits that requires a comprehensive therapeutic approach to be effective at improving self-regulation and everyday function. These deficits can affect a number of critical aspects of individual performance such as awareness, emotional regulation, and self-efficacy. As an alchemy, these serve to be instrumental to TBI patients' emotional regulation capability, and serve as complements to overall satisfactory executive functioning. Efforts have been made in therapeutics to supersede barriers to improving these factors in the form of interventions. Those observed in history had required considerable resources, evident in the apparent high cognitive load and by limits to their effective implementation, wide dissemination and, ultimately, their potential benefit to TBI patients. At present, it is fundamental to explore the benefits of an intervention promising a favorable effect on both attention and present moment awareness (Aim 1), effectiveness in developing emotional regulation and everyday life function (Aim 2), and structured to permit investigation of the functional and structural neural effects on attention (Aim 3). This hypothesis aims to prove these attributes are central to the development of adaptive self-monitoring and self-regulation skills that can be used in a real life environment. The study results will provide valuable information that will ultimately support the refinement of an effective intervention that can have a real impact on patients' ability to improve quality of life, community integration, and supporting an active lifestyle. In addition, acquired neuroimaging will aid in analyzing the effect of the intervention on brain function which will allow for a more established comprehension of the underlying mechanisms driving the benefits, permitting improved design of an effective therapeutic intervention for TBI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of moderate to severe TBI through medical records or interview, based on the Glasgow Coma Scale (GCS) and the definition adopted by the TBI Model Systems National Database (TBIMS NDB), where one of the following criteria must be met:

   * Post traumatic amnesia > 24 hours
   * Trauma related intracranial neuroimaging abnormalities
   * Loss of consciousness exceeding 30 minutes (unless due to sedation or intoxication)
   * GCS in the emergency department of less than 13 (unless due to intubation, sedation, or intoxication);
2. At least 12 months post injury
3. Presence of a deficit in sustained attention as measured by the Attention-Related Cognitive Errors Scale (ARCES) [69] score greater than 3.5 or presence of a deficit in sustained attention as measured by the sustained attention to response task (SART) [64]. Impairment will be defined as having omissions or the reaction time variability scores, two measures of "inattentiveness," one standard deviation above the normative mean.
4. Willingness and ability to participate in all testing and the 10-week intervention and daily home activities/exercises.
5. Medically stable and no plan for major change in medications for at least 6 months or for the duration of the study
6. Have sufficient language functioning to participate in an intervention conducted in English
7. Average memory functioning to be able to benefit from a progression of treatment (as measured by total learning trials on the California Verbal Learning Test-II within 2 standard deviations of the mean)

General Exclusion Criteria:

1. Severe cognitive impairment as defined by a Mini-Mental State Examination score < 18.
2. Any previous neurological injury or illness in addition to the documented TBI (e.g. epilepsy, MS).
3. Active substance abuse
4. Acquired brain injury of nontraumatic origin
5. Be enrolled or currently enrolled in another research study that is likely to affect participation in this research study
6. Significant psychiatric history (e.g. schizophrenia, bipolar disorder) due to the potential influence of such disorders on cognitive functioning (because of the prevalence of depression/anxiety in the TBI population, subjects will not be excluded based on a history of depression/anxiety; rather, these will be controlled by including measures of depression/anxiety as covariates in group-level analyses)
7. Had previously participated in regular mindfulness based activities such as meditation and yoga.

MRI-Specific Exclusion Criteria:

1. Being pregnant or planning to become pregnant
2. Have had a penetrating TBI
3. Left handed (to control for hand dominance effect on neuroimaging)
4. Focal injury if the injury necessitated neurosurgical intervention and/or caused gross derangement of neuroanatomy (Given that TBI is most often represented by mixed pathophysiology and diffuse axonal injury is nearly universal findings, focal injury will not be a systematic exclusionary criteria).
5. For all study participants, additional exclusionary criteria associated with MRI will be discussed and enforced. This includes, conditions contraindicated for MRI (implanted metallic devices-aneurysm clips, pacemakers, claustrophobia for subject safety), surgical hardware in the head or cervical spine will also be excluded due to potential for severe image artifacts. We will be using the RONIC MRI screening form for this purpose.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pre to Post Change in Sustained attention (Response time variability) | Change from pre (baseline) to post (10 weeks) intervention
  Response time variability of the sustained attention to response task (SART) will provide measure of improvement in sustained attention
Pre to Post Change in Sustained attention (commission errors) | Change from pre (baseline) to post (10 weeks) intervention
  Commission errors of the sustained attention to response task (SART) will provide measure of improvement in sustained attention
Pre to Post Change in Present Moment Awareness | Change from pre (baseline) to post (10 weeks) intervention
  Improvement in the ability to attend to the present moment will be measured using the Five Facet Mindfulness Questionnaire (FFMQ). Total score from 1 to 5, higher score representing greater mindfulness
Pre to Post Change in Mindfulness/Present Moment Awareness | Change from pre (baseline) to post (10 weeks) intervention
  Improvement in mindfulness will be measured using the Freiburg Mindfulness Inventory (FMI) Questionnaire. Score ranges between 14 and 56 with higher scores indicating higher mindfulness
Pre to Post Change in Behavioral Measures of Attention | Change from pre (baseline) to post (10 weeks) intervention
  Attention [lapses] will be assessed using the Attention-Related Cognitive Errors Scale (ARCES), as it will provide a measure for the frequency of cognitive failure experiences (i.e. getting distracted, reading without paying attention to content, losing track of a conversation, etc.). Score ranges from 1 to 5 with higher scores indicating greater attention lapses.
Pre to Post Change in Self-Efficacy | Change from pre (baseline) to post (10 weeks) intervention
  Self efficacy will be measured using the Self Efficacy Questionnaire for Symptom Management Scale. Score ranges from 13-130 with higher score indicating greater self-efficacy
Pre to Post Change in Depression | Change from pre (baseline) to post (10 weeks) intervention
  Depression will be measured using the PHQ-8. Score ranges from 0-24 with higher score indicating greater depression.
Pre to Post Change in anxiety | Baseline (1st day); at 10 weeks; following 6 months
  This will be measured using the Spielberger's State Anxiety Inventory (STAI). Score ranges from 20-80, with higher score indicating greater anxiety
Pre to Post Change in emotional regulation | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Difficulty in Emotional Regulation Scale (DERS). Total score ranges from 36-180, with higher score indicating greater problems with emotional regulation.
Pre to Post Change in socio-emotional problem solving | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Social Problem-Solving Inventory - Revised (SPSI-R). Total score ranges from 0-100, with higher score indicating greater social problem-solving ability.

SECONDARY OUTCOMES:
Pre to Post Change in Quality of Life after brain injury | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using Quality of Life After Brain Injury (QOLIBRI).Total score ranges from 0-100, with higher score indicating greater health related quality of life after TBI.
Pre to Post Change in Everyday Function | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using SF12. Total score ranges from 0-100, with higher score indicating greater physical and mental health functioning.
Pre to Post Change in Behavioral Function | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using Functional Behavior Profile. Total score ranges from 0-108, with higher score indicating greater behavioral function.
Pre to Post Change in Awareness | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using Awareness Questionnaire (AQ).Total score ranges from 17-85 with higher score indicating greater function after TBI. Difference scores ( family subtracted from patient ratings) range from -68 to 68, with greater/lower score than 0 associated with greater impaired awareness (rating his function greater/lower than family).
Pre to Post Change in Community Integration | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Community Integration Questionnaire (CIQ). Score ranges from 0 to 29, with higher scores indicating greater independence and community integration.
Pre to Post Change in Socio-emotional behavior executive functioning skills | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Brock Adaptive Functioning Questionnaire. Score ranges from 20 to 100, with lower scores indicating better functioning.
Pre to Post Change in Satisfaction With Life | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using Satisfaction With Life Scale (SWLS). Score ranges from 5-35 with higher score indicating greater life satisfaction.
Pre to Post Change in Emotional Regulation | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Emotional Regulation Questionnaire (ERQ). Items averaged score ranges from 1-7 with higher score indicating greater emotional regulation.
Pre to Post Change in Basic Empathy | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Basic Empathy Scale (BES). Items averaged score ranges from 1-5 with higher score indicating greater empathy.
Pre to Post Change in Empathy Quotient | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Empathy Quotient (EQ). Score ranges from 0-80 with higher score indicating greater empathy.
Pre to Post Change in Neuropsychological Measures - Intelligence | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Wechsler abbreviated scale of intelligence manual (WASI)
Pre to Post Change in Neuropsychological Measures - Verbal learning and memory | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the California Verbal Learning Test (CVLT-II)
Pre to Post Change in Neuropsychological Measures - Processing speed | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Oral Symbol Digit Modalities Test (SDMT)
Pre to Post Change in Neuropsychological Measures - Alertness and Vigilance | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Digit Vigilance Test
Pre to Post Change in Neuropsychological Measures - Attention/executive function | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Paced Auditory Serial Addition Test
Pre to Post Change in Neuropsychological Measures - Executive function in cognitive set shifting and inhibition | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Delis-Kaplan Executive Function System (D-KEFS ) Stroop
Pre to Post Change in Neuropsychological Measures - Executive function in sequential set-shifting | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Oral Trail Making Test
Pre to Post Change in Neuropsychological Measures in Executive function - Verbal Fluency | Change from pre (baseline) to post (10 weeks) intervention
  This will be measured using the Delis-Kaplan Executive Function System (D-KEFS ) Verbal Fluency

CONTACTS AND LOCATIONS:
Overall Officials: Jean Lengenfelder, Ph.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States